CLINICAL TRIAL: NCT04242134
Title: Comparison of Noncompliant Balloon With Drug-coating Balloon Angioplasties for Side Branch After Provisional Stenting for Patients With True Coronary Bifurcation Lesions
Brief Title: Drug-coating Balloon Angioplasties for True Coronary Bifurcation Lesions
Acronym: DCB-BIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20191128
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1 randomization to either PS-DCB which will be the treatment group or PS-NCB which will be the control group based on an online Clinical Research Data Management Platform provided by King Yee, Beijing CN. The initiation of the trial is defined as the time of randomization. After study subjects' enrollment and randomization, the study intervention will take place immediately. The follow-up visits for the primary endpoint are scheduled at 1, 6, and 12 months after the index procedure. Angiographic follow-up is scheduled at 13 months.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will remain blinded until the final study results are released.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS-DCB (Experimental): For PS-DCB group
  1. NC balloon dilating ostial side branch (SB) (1:1 ratio).
  2. DCB dilating SB. Specifically, the DCB, which had to be 2-3 mm longer on each side than the predilatation balloon, was inflated at nominal pressure for 30~ 60 s. The ratio of the DCB diameter to the nominal diameter of the SB was recommended to be between 0.8 and 1.0. DCB should be delivered to the lesion within 2 min after entering human body.
  3. Kissing inflation using 2 noncomplian balloons.
  4. Stenting side branch with T and protrusion (TAP) technique if any of the following issues was observed after kissing balloon inflation: >type C dissection or thrombolysis in myocardial infarction (TIMI) flow <3.
  5. Final kissing inflation and proximal optimal technique (POT).
  Interventions: Device: Drug-coating balloon
- PS-NCB (Active Comparator): For PS-NCB group
  1. NC balloon dilating ostial SB (1:1 ratio).
  2. Kissing inflation using 2 NC balloons.
  3. Stenting side branch with TAP technique if any of the following issues was observed after kissing balloon inflation: >type C dissection or thrombolysis in myocardial infarction (TIMI) flow <3.
  4. Final kissing inflation and proximal optimal technique (POT).
  Interventions: Device: Drug-coating balloon

INTERVENTIONS:
Device: Drug-coating balloon — Provisional stenting technique with DCB
  Other Names: DCB

SUMMARY:
This study is designed to investigate whether drug-coated balloon (DCB) compared to conventional balloon angioplasty for side branch after provisional stenting will lead to lower rates of the composite endpoint of major adverse cardiac event (MACE) at 12 months. The individual components of MACE include cardiac death, myocardial infarction (MI), or target lesion revascularization (TLR). True bifurcation lesions were defined according to Medina classification.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized-controlled, single blind, superiority trial that will include 25 international sites. The investigators aim to enroll 784 subjects with true coronary bifurcation lesions in native coronary arterial segments.

All patients with true coronary bifurcation lesions suitable for angioplasty will undergo 1:1 randomization either to PS (provisional stenting)-DCB or PS-NCB (noncompliant balloon) group using a randomization schedule blocked by site.

All subjects will be screened according to the predefined inclusion and exclusion criteria per protocol and will further undergo angiography after successful stenting of the main vessel with ostium side branch visually estimated stenosis ≥70%. Data and images will be collected during the index procedure, during re-intervention in the case of clinically driven revascularization, and at the predefined 12-month clinical follow-up visit. All subjects will also undergo angiographic follow-up at 13 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be age ≥18 years.
2. Subject has silent ischemia, or stable/unstable angina, or acute MI older than 1-week from the onset of chest pain to admission.
3. Subject (or legal guardian) understands the trial design and treatment procedures and provides written informal consent before any trial-specific tests or procedures are performed.
4. Subject is willing to comply with all protocol-required follow-up evaluations.
5. Target lesion must be a true bifurcation lesion on coronary angiography (defined as Medina 0,1,1, Medina 1,0,1, or Medina 1,1,1 coronary bifurcation lesions) and is eligible for percutaneous coronary intervention (PCI).
6. Target lesion reference vessel diameter (both main vessel and side branch) ≥ 2.5 mm by visual estimation.
7. Target lesion must have visually estimated stenosis ≥50%.
8. Target lesion length of side branch must be <10 mm by visual estimation.
9. Ostium side branch must have visually estimated stenosis ≥70% after stenting of the main vessel.

Exclusion Criteria:

1. Patient with STEMI (within 1-week from the onset of chest pain to admission).
2. Patient has known allergy to the study balloon/stent system or protocol-required concomitant medications.
3. Patient is intolerable to dual anti-platelet therapy.
4. Patient has any other serious medical illness that may reduce life expectancy to less than 12 months.
5. Patient is pregnant or nursing.
6. Patient is participating in another clinical trial that has not reached its primary endpoint within 24 months after the index procedure.
7. Patient has a planned procedure that may cause non-compliance with the protocol or confound data interpretation.
8. Restenotic lesion.
9. Chronic total occlusion (CTO) lesion in either main vessel or side branch is not successfully recanalized.
10. Severe calcification needing rotational atherectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac event | 12 months after angioplasty
  MACE defined as the composite of cardiac death, myocardial infarction (MI), and clinically driven TLR.

SECONDARY OUTCOMES:
Rate of all-cause death or cardiac death | 12 months after angioplasty
  In general, all deaths are considered cardiac unless an alternate cause is unequivocally established, even among subjects with serious noncardiac comorbidities.
Rate of periprocedural MI, Spontaneous MI, or target vessel MI | 12 months after angioplasty
  According to the DCB-BIF trial definition.
Rate of clinically-driven TLR or TVR | 12 months after angioplasty
  Clinically driven revascularization includes repeat PCI or coronary artery bypass graft (CABG) for recurrent or persistent symptomatic ischemia and can be defined according to the relationship to the index PCI (target lesion).
Rate of thrombosis | 12 months after angioplasty
  The safety endpoint was stent thrombosis (ST), according to the definition by Academic Research Consortium.

OTHER OUTCOMES:
Rate of Angiographic success | 1 day
  PCI is considered successful for lesions treated with stent implantation if the residual diameter stenosis based on visual estimation is less than or equal to 10% and the final TIMI flow grade is 3. PCI is considered successful for lesions treated without stent implantation if the residual diameter stenosis based on visual estimation is less than or equal to 20% and the final TIMI flow grade is 3.
Rate of clinical procedural success | 7 day
  Successful PCI without MACE during hospital stay.
Crossover rate | 1 day
  From single stent technique to two-stent technique

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao XF, Ge Z, Kan J, Kong XQ, Wang Y, Qiu CG, Tresukosol D, He YQ, Wu Q, Li JF, Yuan HT, Shen C, Chen X, Munawar M, Hanif B, Santoso T, Shin ES, Sheiban I, Ye F, Zhang JJ, Chen SL; DCB-BIF investigators. Rationale and design for comparison of non-compliant balloon with drug-coating balloon angioplasty for side branch after provisional stenting for patients with true coronary bifurcation lesions: a prospective, multicentre and randomised DCB-BIF trial. BMJ Open. 2022 Mar 11;12(3):e052788. doi: 10.1136/bmjopen-2021-052788. PMID 35277400